CLINICAL TRIAL: NCT03206840
Title: The Neural Correlates of the " Self " in Altered States of Consciousness
Brief Title: Neural Correlates of Self
Acronym: NeuCoSe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL17_0274; 2017-A01923-50 (Other: ID-RCB)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: mindfulness meditation; hypnosis; meta-awareness; absorption; consciousness; self
MeSH Terms: interventions — Meditation; Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): three instructions will be given to each participant: "control", "meditation", "hypnosis". The order of "meditation" and "hypnosis" will be randomized amongst two groups to avoid order effects.
  Interventions: Behavioral: "control", "meditation", "hypnosis".
- Group 2 (Experimental): three instructions will be given to each participant: "control", "meditation", "hypnosis". The order of "meditation" and "hypnosis" will be randomized amongst two groups to avoid order effects.
  Interventions: Behavioral: "control", "meditation", "hypnosis".

INTERVENTIONS:
Behavioral: "control", "meditation", "hypnosis". — three instructions will be given to each participant: "control", "meditation", "hypnosis". The order of "meditation" and "hypnosis" will be randomized amongst two groups to avoid order effects.

SUMMARY:
Despite the increasing popularity of mindfulness meditation and hypnosis in healthcare and in the general community the underlying neurobiological mechanisms are unclear. The change in the relationship between the self and the conscious experience that they bring about may be crucial. This study aims to identify the neural correlates of self-consciousness in meta-awareness and absorption - using functional Magnetic Resonance Imaging (fMRI) in healthy participants combined with detailed first-person experiential accounts and behavioural tasks. This study will provide important clues about the widely reported effects of mindfulness meditation and hypnosis and shed light on the neural correlates of the conscious experience of self.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70
* Body mass index between 18.5 and 30
* Covered by health insurance
* motivated to participate
* signed informed consent
* normal or corrected-to-normal eyesight
* sufficient command of French to be able to follow the instructions

Exclusion Criteria:

* history of neurological or psychiatric conditions
* chronic pain or another medical condition altering pain perception
* use of medication that affects the central nervous system
* use of opioids or antidepressant medication
* severe auditory loss
* consumption of alcohol or intoxicants on the day of the experiments and the day preceding the experiments
* pregnancy, breastfeeding or having given birth <6months ago
* any contra-indication to Magnetic Resonance Imaging (metal implants or foreign bodies), agitation, claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Reaction time (minutes) | at day 1
  reaction times during behavioural tasks.
Brain activation with IRM | At day 3
  Activation of different brain areas, as measured with functional Magnetic Resonance

SECONDARY OUTCOMES:
personality trait with questionnaires | at day 2
  scores on different personality questionnaires
Scores during behavioural tasks | at day 1
  scores on likert scale (1-5 and 1-9) about intensity of the stimui presented during the task
Scores during behavioural tasks | at day 3
  scores on likert scale (1-5 and 1-9) about intensity of the stimui presented during the task
salivary volume (millimeter) | at day 1
  salivary volume after behavioural tasks

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LUTZ, PhD, Principal Investigator — Lyon Neuroscience Research Center
Locations (1):
- Hospices Civils de Lyon Hôpital le Vinatier/Inserm, Bron, France

REFERENCES:
- [Result] Lutz A. Regulation of attention and emotions by meditation: neurophysiological basis and implications for mental and physical health. In: 12th BIAL Foundation Symposium "Amplified states of consciousness"; 2018 Apr 6; Porto, Portugal. Lutz A. Méditation, hypnose… se soigner par la conscience. In: INSERM - Culture scientifique (webinar); 2022 Dec 13; Paris, France (online). Lutz A. Mindfulness meditation from the lenses of phenomenology and neurosciences. In: USC Center for Mindful Science - Invited lecture; 2022 Dec 12; Los Angeles (CA), USA. Lutz A. Neurophenomenology after Varela (1996). In: Metanoia/Ouroboros - Seminar; 2021 Sep 1; (online).